CLINICAL TRIAL: NCT07164729
Title: Comparison of the Effects of Dynamic and PNF Stretching Applied to the Quadriceps Muscle Group on Muscle Performance, Muscle Strength, and Joint Range of Motion in Professional Cyclists
Brief Title: Dynamic vs. PNF Quadriceps Stretching in Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 02092025
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sports Physical Therapy
Keywords: Cycling; Sports; Power; Jumping; Anaerobic Performance
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Stretching (Experimental)
  Interventions: Other: PNF Stretching
- Dynamic Stretching (Experimental)
  Interventions: Other: Dynamic Stretching

INTERVENTIONS:
Other: PNF Stretching — Dynamic stretching of the quadriceps will be performed using walking lunges. This exercise dynamically stretches the quadriceps and hip flexors while also improving balance and coordination. During the exercise, participants stand upright, step one leg forward, and lower their body by bending the knee. They then step forward with the other leg to complete the movement. Ten steps will be performed for each leg.
  Arms: PNF Stretching
Other: Dynamic Stretching — The "Hold-Relax" technique will be applied. Hold-Relax PNF stretching is based on the principle of isometric contraction of the muscle followed by passive stretching. This technique is effective for increasing muscle flexibility and reducing muscle tension. The medial and lateral parts of the quadriceps will be stretched by Flexion-Adduction-External Rotation and Flexion-Abduction-Internal Rotation patterns3. During the exercise, participants will lie prone with the knee flexed. They will be asked to attempt knee extension while the movement is resisted by the physiotherapist. The contraction will be maintained for 10 seconds, after which the participant will be instructed to relax. Following relaxation, the knee flexion angle will be increased. Ten repetitions will be performed for each leg.
  Arms: Dynamic Stretching

SUMMARY:
Following an initial assessment, 30 professional cyclists will be divided into two groups (1:1). PNF stretching will be applied to the Quadriceps muscles of the participants in Group A, while Group B will perform dynamic stretching on the Quadriceps muscles. After the interventions, all participants will undergo a second assessment. The study aims to compare the immediate effects of these two different types of stretching on muscle performance, strength and joint range of motion. Participants will attend a single day for both the assessments and the intervention sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being a professional cyclist (training intensively at least 4-5 times per week and having a minimum of 5-10 years of cycling experience).
* Voluntary participation in the study.
* No recent history of sports-related injury.

Exclusion Criteria:

* Presence of neurological, orthopedic, or cardiovascular diseases.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Test | Through study completion, an average of 1 month
  The vertical jump test is performed by instructing an athlete to jump as high as possible from a standing position. Typically, the athlete will first stand and reach upward to mark the highest point they can touch while standing. Then, they will jump as high as possible, and the jump height will be recorded. The difference between the standing reach and jump height is calculated as the vertical jump distance.
Anaerobic Power Step Test | Through study completion, an average of 1 month
  It involves stepping up and down on a platform of a specified height. The participant will step rapidly and rhythmically on the platform for 30 and 60 seconds, aiming to complete as many steps as possible. The total number of steps will be recorded at the end of the test. Proper form and rhythmic stepping will be emphasized during the test; the athlete must place the entire foot on the platform and achieve full extension with each step. The data obtained from this test will be used to assess the athlete's anaerobic capacity and lower-body explosive power

SECONDARY OUTCOMES:
Lower Extremity Muscle Strength | Through study completion, an average of 1 month
  Lower extremity muscle strength will be measured using the Lafayette Hand-Held Dynamometer (HHD). During its application, the Lafayette HHD measures the force generated during the muscle's maximal isometric contraction. Knee flexion, knee extension, hip flexion and hip extension muscle strength will be measured. The measurement will be repeated three times.
Lower Extremity Joint Range of Motion | Through study completion, an average of 1 month
  Lower extremity joint range of motion will be assessed using a goniometer. The joint range of motion measurements will include hip flexion, extension, abduction, adduction, internal and external rotation, as well as knee flexion and extension.

CONTACTS AND LOCATIONS:
Overall Officials: Çiçek Günday, Asst. Prof., Principal Investigator — Istinye University; Arda Akça, Physiotherapist, Study Chair — Istinye University; Elif Berfin Bulut, Physiotherapist, Study Chair — Istinye University
Locations (1):
- Istinye University Physiotherapy and Rehabilitation Application and Research Center (İSÜFİZYOTEM), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No